CLINICAL TRIAL: NCT00117247
Title: A Study to Assess the Pharmacokinetics and Pharmacodynamics of Repeat-Sose Subcutaneous Darbepoetin Alfa in Subjects With Congestive Heart Failure and Anemia, and a Single Dose in Healthy Age- and Sex-Matched Control Subjects
Brief Title: A Study of Repeat-Dose Subcutaneous Darbepoetin Alfa in Subjects With Congestive Heart Failure and Anemia, and a Single Dose in Healthy Age- and Sex-Matched Control Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20010198
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Anemia; Congestive Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Anemia; Heart Failure | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The purpose of this study is to evaluate the single dose pharmacokinetics (PK) of subcutaneous (SC) darbepoetin alfa in subjects with congestive heart failure (CHF) and anemia.

ELIGIBILITY:
Inclusion Criteria: - Symptomatic CHF despite optimized therapy for at least the previous 3 months (treatment included a diuretic, angiotensin converting enzyme [ACE] inhibitor, and/or an A2 antagonist, unless not tolerated) - Hemoglobin greater than or equal to 12.5 g/dL at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2004-07

PRIMARY OUTCOMES:
Pharmacokinetic profiling of Aranesp® in HF pts

SECONDARY OUTCOMES:
Pharmacodynamic responses (hgb) following Aranesp® administration in HF patients

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com